CLINICAL TRIAL: NCT02025062
Title: Impact of Comprehensive Geriatric Assessment on Malnutrition, Functional Status and Survival in Elderly Patients With Head and Neck Squamous Cell Carcinomas (HNSCCs): a Randomized Controlled Multicenter Clinical Trial
Brief Title: Comprehensive Geriatric Assessment and Head and Neck Elderly Cancer Patients
Acronym: EGéSOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cancéropole Ile De France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K120902; 2013-A00437-38 (Other: NCI)
Record Dates: First submitted 2013-11-21; First posted 2013-12-31 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Head and Neck Squamous Cell Carcinomas (HNSCCs)
Keywords: head and neck squamous cell carcinomas (HNSCCs); elderly; cancer; comprehensive geriatric assessment; functional status; malnutrition; survival
MeSH Terms: conditions — Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): In the control arm, patients are followed-up by the head-and-neck physician, oncologist and radiotherapists and did not benefit of Comprehensive Geriatric Assessment.
- Comprehensive Geriatric Assessment (Experimental): The CGA (Comprehensive Geriatric Assessment) is a multidimensional assessment of general health status, using validated scales. It produces an inventory of problems which can then serve to develop an individualized geriatric intervention plan of care and follow-up.
  Interventions: Other: CGA and geriatric follow-up

INTERVENTIONS:
Other: CGA and geriatric follow-up — The CGA is a multidimensional assessment of general health status, using validated scales. It produces an inventory of problems which can then serve to develop an individualized geriatric intervention plan of care and follow-up
  Arms: Comprehensive Geriatric Assessment

SUMMARY:
The intervention tested in this research project aims to reduce this inequality by improving the management of elderly head and neck cancer patients with a specific management. Indeed, the treatment of elderly head and neck cancer patients has specificities concerning treatment options, their tolerance, psychological management, nutritional and functional status, and support needed at home. To assess the overall needs of the elderly patients, an assessment known as "comprehensive geriatric assessment" (CGA) can be performed by a geriatrician with extensive testing and questionnaires. This assessment is long and requires an experienced geriatrician. It leads to the development of an individualized treatment plan (physiotherapy, psychological follow-up, support at home, nutritional management ...) and follow-up to adapt the necessary cares for the duration of the cancer treatment. The CGA utility has been studied in elderly patients with nonmalignant diseases. Studies have shown that CGA allowed improving survival and maintaining the elderly at home.

DETAILED DESCRIPTION:
Context: The survival of elderly patients with head and neck squamous cell carcinomas (HNSCC) cancer is greatly reduced compared to younger subjects. Several explanations have been proposed : a competitive comorbidity, a more frequent refusal of standard therapy or the choice of a suboptimal treatment due to fear of toxicities. The comprehensive geriatric assessment (CGA) may influence the decision-making process and help for managing elderly patients with head and neck cancer. The CGA is a multidimensional assessment of general health status, using validated scales. It produces an inventory of problems which can then serve to develop an individualized geriatric intervention plan of care and follow-up.

Hypotheses: We postulate that the CGA and the geriatric follow-up improves 1) the therapeutic decision-making process thanks to a better assessment of the patient's functional reserve and its capacity to support or not the treatment, and 2) the overall survival, the functional status and the nutritional status of elderly patients with HNSCC because of a more appropriate treatment and a personalized medical follow-up after surgery and/or radiotherapy and/or chemotherapy or more rarely targeted therapy, with adjustment of treatments and management of comorbidities and/or treatment complications.

Main objective: To assess the impact of the CGA and the geriatric follow-up on the overall survival, the functional status and the nutritional status of elderly patients with HNSCC.

Secondary objectives: To assess the impact of the CGA on the therapeutic decision, the toxicity and/or complications of treatment, the complete realization of treatment, the autonomy, the institutionalization, the total hospitalization stay, the quality of life of elderly patients with HNSCCs and the costs.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 years old and over (modified by amendment n 2 -1/07/2014)
* macroscopical lesions suggesting an cancerous tumor in head and neck awaiting pathology confirmation;
* support in one of ENT/Maxilla-facial surgery departments in the study;
* patients insured by a social security;
* patients informed of the study, and having given his non opposition verbally.

Exclusion Criteria:

* patients deprived of liberty or under legal protection;
* presence of psychological, family, socials or geographic condition(s) that may interfere with the proper conduct of the study;
* personal history of head and neck cancer except single surgery for squamos cell carcinoma without additional treatment (without curietherapy or RT) with a free interval of at least 5 years (modified by amendment n 2 -1/07/2014)
* patients with cancerous tumor of sinus and salivary glands

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 499 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Composite criteria, including: death; autonomy (if loss of two points or more in the Activity of Daily Living (ADL) compared with the initial ADL); nutritional status (if weight loss of 10% or more compared to the initial weight at diagnosis | 6 months after the randomization

SECONDARY OUTCOMES:
progression-free survival | 6 month, 12 month and 24 month after the randomization
death | 6 month , 12 month and 24 month after the randomization
total duration of hospitalization | 6 month, 12 month and 24 month after the randomization
quality of life (QLQC30, HN35) | 6 month , 12 month and 24 month after the randomization
costs of treatment | 6 month , 12 month and 24 month after the randomization

CONTACTS AND LOCATIONS:
Overall Officials: Eléna Paillaud, MD / PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Lydia Brugel, MD / PhD, Principal Investigator — Centre Hospitalier intercommunal de Créteil
Locations (1):
- Centre Hospitalier Intercommunal de Créteil / Hopital Henri Mondor, Créteil, France

REFERENCES:
- [Background] Abstracts of the 6th European Congress of Oto-Rhino-Laryngology Head and Neck Surgery, June 30-July 4, 2007, Vienna, Austria. Eur Arch Otorhinolaryngol. 2007 Jun;264 Suppl 1:S1-354. doi: 10.1007/s00405-007-0343-8. No abstract available. PMID 17558509
- [Background] Homma A, Sakashita T, Oridate N, Suzuki F, Suzuki S, Hatakeyama H, Mizumachi T, Taki S, Fukuda S. Importance of comorbidity in hypopharyngeal cancer. Head Neck. 2010 Feb;32(2):148-53. doi: 10.1002/hed.21158. PMID 19536763
- [Derived] Lafont C, Paillaud E, Bertolus C, Baron M, Caillet P, Bouvard E, Laurent M, Salvan D, Chaumette L, de Decker L, Piot B, Barry B, Raynaud-Simon A, Sauvaget E, Minard A, Anota A, Panjo H, Brugel L, Canoui-Poitrine F. Geriatric assessment and quality of life for 2 years in older patients with head and neck cancer. J Natl Cancer Inst. 2024 May 8;116(5):758-763. doi: 10.1093/jnci/djae027. PMID 38335935
- [Derived] Brugel L, Laurent M, Caillet P, Radenne A, Durand-Zaleski I, Martin M, Baron M, de Kermadec H, Bastuji-Garin S, Canoui-Poitrine F, Paillaud E. Impact of comprehensive geriatric assessment on survival, function, and nutritional status in elderly patients with head and neck cancer: protocol for a multicentre randomised controlled trial (EGeSOR). BMC Cancer. 2014 Jun 13;14:427. doi: 10.1186/1471-2407-14-427. PMID 24923533